CLINICAL TRIAL: NCT05404945
Title: Fitness-adapted, Pembrolizumab-based Therapy for Untreated Classical Hodgkin Lymphoma Patients 60 Years of Age and Above (cHL 001)
Brief Title: Fitness-adapted, Pembrolizumab-based Therapy for Untreated Classical Hodgkin Lymphoma Patients 60 Years of Age and Above
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University of Virginia (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Principal Investigator, Craig A Portell, MD, Associate Professor of Medicine, University of Virginia
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: cHL001
Record Dates: First submitted 2022-05-22; First posted 2022-06-03 (Actual); Last update posted 2024-07-03 (Actual); Status verified 2024-06

CONDITIONS: Classical Hodgkin Lymphoma
MeSH Terms: interventions — pembrolizumab; Doxorubicin; Vinblastine; Dacarbazine; Brentuximab Vedotin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Fit Cohort (Experimental): Three 6-week cycles of 400 mg intravenous pembrolizumab + intravenous AVD (q 2 weeks).
  Interventions: Drug: Pembrolizumab; Drug: Doxorubicin; Drug: Vinblastine; Drug: Dacarbazine; Drug: Brentuximab vedotin
- Frail Cohort (Active Comparator): Three 6-week cycles of 400 mg intravenous pembrolizumab and concurrent (q 3 week) intravenous brentuximab vedotin (BV).
  Interventions: Drug: Pembrolizumab; Drug: Doxorubicin; Drug: Vinblastine; Drug: Dacarbazine; Drug: Brentuximab vedotin
- Unfit Cohort (Active Comparator): Three 6-week cycles of 400 mg intravenous pembrolizumab and mini-AVD (q 2 weeks).
  Interventions: Drug: Pembrolizumab; Drug: Doxorubicin; Drug: Vinblastine; Drug: Dacarbazine; Drug: Brentuximab vedotin

INTERVENTIONS:
Drug: Pembrolizumab — Pembrolizumab 400 mg IV
Drug: Doxorubicin — Doxorubicin 25mg/m2 IV
  Other Names: Adriamycin
Drug: Vinblastine — Vinblastine 6mg/m2 IV
Drug: Dacarbazine — Dacarbazine 375mg/m2 IV
Drug: Brentuximab vedotin — Brentuximab vedotin 1.8 mg/kg IV

SUMMARY:
This is a multi-center, open-label phase II study to assess the efficacy of a novel fitness-adapted regimen in previously untreated older patients with classical Hodgkin lymphoma. All participants will receive up to a total of 8 cycles of pembrolizumab (Q6 week dosing). The first cycle of pembrolizumab will be administered in combination with brentuximab vedotin (BV) ("lead-in treatment").

Following lead-in treatment, all participants will undergo interim PET/CT (iPET) as well as fitness testing to help inform participant level of fitness for subsequent lymphoma-directed therapies.

Participants deemed "Frail" by this assessment will continue 3 additional 6 week cycles of concurrent pembrolizumab and BV ("induction therapy", each cycle is 42 days), then continue single-agent pembrolizumab to complete up to 4 additional cycles (i.e., 8 total) of therapy ("consolidation and maintenance therapy", Frail cohort). Two additional BV doses will be given as consolidation, at days 1 and 22 of pembrolizumab cycle 5.

Those deemed "fit" after lead-in therapy (Fit cohort) will continue pembrolizumab and switch from BV to concurrently-administered combination chemotherapy using doxorubicin (A), vinblastine (V), and dacarbazine (D) for a total of 4 planned AVD cycles (3, 6-week pembrolizumab cycles, "induction therapy"). Chemotherapy drugs will be given at standard doses as in ABVD (no bleomycin will be given in this study) on days 1 and 15 of each 28-day cycle (C1AVD), and pembrolizumab dosing will remain every 42 days. Following end-induction PET/CT, pembrolizumab will continue every 42 days for up to 4 cycles in the consolidation/maintenance phase. Two additional BV doses will be given as consolidation, at days 1 and 22 of pembrolizumab cycle 5.

Participants deemed "unfit" after lead-in therapy and by fitness assessment will continue pembrolizumab and switch from BV to concurrently administered combination chemotherapy termed "mini-avd" as induction therapy. Mini-avd consists of lower doses of conventional AVD chemotherapy (doxorubicin, vinblastine and dacarbazine) and will be administered for on days 1 and 15 of a 28 day cycle for 4 planned cycles. Pembrolizumab will continue every 42 days. Following end-induction PET/CT, pembrolizumab will continue every 42 days for up to 4 cycles in the consolidation/maintenance phase. Two additional BV doses will be given as consolidation, at days 1 and 22 of pembrolizumab cycle 5.

ELIGIBILITY:
Inclusion Criteria:

* Participants of any sex who are ≥60 years of age on day 1, cycle 1.
* The participant must be willing and able to provide written informed consent for the trial and participate in all planned study procedures.
* Histologically confirmed diagnosis of classical Hodgkin lymphoma
* PET-avid, measurable disease (≥1.5cm bi-dimensional measurement)
* Have an Eastern Cooperative Oncology Group (ECOG) performance status (PS) of 0 to
* PS 2 may be allowed at the discretion of the treating investigator if impairment is considered to be primarily lymphoma-related. Evaluation of ECOG is to be performed within 10 days prior to the date of registration.
* Participants who have received involved field radiation will be allowed. However, they will be excluded if any of the following are true:

  1. Radiation was dosed ≤6 months from registration.
  2. Radiation was delivered to > 1 lymph node group as defined by the NCCN criteria.
  3. The radiation dose was ≥30 Gy.
  4. The participant has radiation-related toxicities ≥ Grade 2 at the time of registration.
  5. The participant requires corticosteroids for radiation-related toxicities at the time of registration (regardless of dose).
  6. The participant has ever experienced radiation pneumonitis.
* Have adequate organ function as defined per protocol. Specimens must be collected within 10 days prior to registration (confirmation of eligibility).

Exclusion Criteria:

* Nodular lymphocyte-predominant Hodgkin lymphoma
* Life expectancy < 6 months for any reason excluding lymphoma
* Has received prior therapy with an immune checkpoint inhibitor, against targets including but not limited to PD1, PDL1, PDL2, CTLA-4, OX40, or LAG 3 unless given with curative intent for reasons other than lymphoma AND the last dose was more than 3 years from registration. Any participant who received prior immune checkpoint inhibitor therapy will be excluded if they experienced any toxicity related to or possibly related to the immunotherapy that required discontinuation of drug.
* Prior systemic therapy for cHL, with the exception of steroids
* If participant received major surgery, they must have recovered adequately from the toxicity and/or complications from the intervention prior to starting study treatment.
* Presence of Grade ≥ 2 sensory and/or motor neuropathy
* Prior solid organ or stem cell transplant.
* Clinical suspicion or evidence of active involvement of lymphoma into the spinal cord, cerebral spinal fluid, or brain. External compression of the spinal cord or nerve roots is not considered involvement.

Has received a live vaccine or live-attenuated vaccine within 30 days prior to the first dose of study drug. Administration of killed vaccines, subunit vaccines, and nucleic acid vaccines is allowed.

* Is currently participating in or has participated in a study of an investigational agent or has used an investigational device within 4 weeks prior to the first dose of study treatment.

Note: Participants who have entered the follow-up phase of an investigational study may participate as long as it has been 4 weeks after the last dose of the previous investigational agent.

* Has a diagnosis of immunodeficiency or is receiving chronic systemic steroid therapy (in dosing exceeding 10 mg daily of prednisone equivalent [excluding steroids needed for lymphoma related symptoms]) or any other form of immunosuppressive therapy within 7 days prior to the first dose of study drug.
* Known additional malignancy that is progressing or has required active treatment within the past 3 years. Note: Participants with basal cell carcinoma of the skin, squamous cell carcinoma of the skin or carcinoma in situ (excluding carcinoma in situ of the bladder) that have undergone potentially curative therapy are not excluded.
* Has known severe hypersensitivity (≥Grade 3) to pembrolizumab and/or any of its excipients.
* Has active autoimmune disease that has required systemic treatment in the past 2 years (i.e. with use of disease modifying agents, corticosteroids or immunosuppressive drugs). Replacement therapy (eg., thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, etc.) is not considered a form of systemic treatment.
* Interstitial lung disease or a history of (non-infectious) pneumonitis/interstitial lung disease that required steroids or has current pneumonitis/interstitial lung disease.
* Any known history of pancreatitis as defined by Gandhi et al. 201432,36.
* Has an active infection requiring oral or intravenous systemic therapy.
* Has a known history of Human Immunodeficiency Virus (HIV).
* Has a known history of Hepatitis B (defined as Hepatitis B surface antigen [HBsAg] reactive) or known active Hepatitis C virus (defined as HCV RNA [qualitative] is detected) infection. Prior exposure to hepatitis B is allowed as long as there are no HBsAg detected (ie positive Hepatitis B core antibody with negative HBsAg). Prior treatment with Hepatitis C is allowed if the screening HCV RNA by PCR is negative.
* Has a known history of active tuberculosis (TB; Mycobacterium tuberculosis).
* Is currently taking a strong CYP3A4 modulator. Subjects taking strong CYP34A modulators that can safely stop these medications prior to treatment should complete a washout period of 4 weeks or 5 times the half-life of a particular drug, whichever is shorter.
* Has a history or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the study, interfere with the participant's participation for the full duration of the study, or is not in the best interest of the participant to participate, in the opinion of the treating investigator.
* Has known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial.
* Is pregnant or breastfeeding, or expecting to conceive or father children within the projected duration of the study, starting with the screening visit through 120 days after the last dose of trial treatment.

Note: given older age at enrollment, WOCBP are not anticipated to enroll on this study.

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Estimated)
Dates: Start 2022-07-26 (Actual); Primary Completion 2027-10-03 (Estimated); Study Completion 2027-10-03 (Estimated)

PRIMARY OUTCOMES:
Complete Remission Rate | 2 years
  Evaluate complete remission rate as defined by LYRIC criteria at end of induction in fit and unfit older participants with cHL following anthracycline-based chemotherapy.
Incidence of grade 3-5 treatment-related AEs | 2 years
  Assess tolerance and safety of a fitness-adapted pembrolizumab-based regimen in fit older participants with cHL based on incidence of grade 3-5 treatment-related AEs (CTCAE v5.0)

SECONDARY OUTCOMES:
2-year PFS, 2-year OS, 2-year Lymphoma Specific Survival in the fit older population following pembrolizumab-based adaptive therapy | 2 years
  Evaluate the efficacy, as determined by the 2-year progression free survival (PFS), overall survival (OS), and 2-year lymphoma specific survival in the fit older population.
Complete remission rate (by LYRIC criteria), 2-year PFS, 2-year OS, 2-year Lymphoma Specific Survival in the Frail older population | 2 years
  Evaluate the efficacy of a chemotherapy-free approach (pembrolizumab plus BV), as determined by the complete remission rate (LYRIC criteria), 2-year progression free survival (PFS), overall survival (OS), and 2-year lymphoma specific survival in participants who are not frail for anthracycline-based therapy.
Complete remission rate (LYRIC criteria) after lead-in BV/pembrolizumab | 2 years
  Assess the efficacy of short course lead-in therapy and correlation with end-induction treatment efficacy for all participants.
Incidence of grade 2-5 immune-related toxicities (CTCAE v5.0) | 2 years
  Assess safety, as determined by the frequency of higher-grade immune-related adverse events for all participants.

OTHER OUTCOMES:
Rate of Indeterminate Response (LYRIC criteria) | 2 years
  Assess the rate of "indeterminate response" by LYRIC criteria at interim and end-induction PET/CT and correlate with the presence of active Hodgkin lymphoma on biopsy (when available) and clinical outcome for all participants.
Incidence of change in fitness assignment from baseline assessment. | 2 years
  Evaluate and summarize incidence of changes in fitness assignments throughout therapy.
Incidence and Severity of treatment-related toxicities | 2 years
  Summarize participant fitness throughout therapy by incidence and severity of treatment-related toxicities.

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - Rutgers Cancer Institute of New Jersey, New Brunswick, New Jersey
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - University of Virginia, Charlottesville, Virginia

IPD SHARING:
Plan to Share IPD: No